CLINICAL TRIAL: NCT04109274
Title: Evaluation of a Novel Strategy to Implement Exercise Evidence Into Clinical Practice in Breast Cancer Care: The NEXT-BRCA Trial
Brief Title: Implementing Exercise Into Clinical Practice in Breast Cancer Care
Acronym: NEXT-BRCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NEXT-BRCA
Record Dates: First submitted 2019-09-05; First posted 2019-09-30 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: exercise; physical activity; self-management
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise; Self-Management

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Institution-Based Exercise and Self-Management (EXSM) (Experimental): Eight session of supervised exercise within the cancer institution plus 8 self-management modules focusing on goal setting and action planning for safe and effective exercise strategies (this is based on our team's successful pilot intervention). Four booster sessions will be provided to this group.
  Interventions: Behavioral: Exercise; Behavioral: Self-Management; Behavioral: Booster Sessions
- Institution-Based Self-management only (SM) (Experimental): Eight SM sessions for safe and effective exercise strategies will be provided to this group (described above). Four booster sessions will be provided to this group.
  Interventions: Behavioral: Self-Management; Behavioral: Booster Sessions
- Usual care (No Intervention): Participants in this group will receive care as normally provided by their treating oncologist. This can be heterogeneous between different physicians and centres, but usually includes oncologists encouraging their patients to 'stay active'

INTERVENTIONS:
Behavioral: Exercise — Exercise component: Aerobic exercise, using recumbent bikes, delivered within the cancer institution. Participants will take part in up to 30-minutes of moderate intensity (50-70% HRmax or 4-6/10 on Rate of Perceived Exertion scale)6 exercise for eight sessions during chemotherapy. An exercise specialist with experience in cancer rehabilitation will supervise the exercise component.
  Other Names: Physical Activity; self-management
  Arms: Institution-Based Exercise and Self-Management (EXSM)
Behavioral: Self-Management — Eight SM modules will be delivered to participants. They will be viewed on an iPad prior to or after the exercise component. The goal of these modules is to aid participants in developing physical activity goals and action plans to continue with between sessions, with an overarching goal of helping them reach exercise guidelines for cancer survivors and the Canadian Physical Activity Guidelines
  Arms: Institution-Based Exercise and Self-Management (EXSM); Institution-Based Self-management only (SM)
Behavioral: Booster Sessions — Four booster sessions will be provided to participants in this group. These will occur at 2, 4, 6, and 8 months post intervention completion. An assessor trained in behavioural counselling will provide booster sessions by phone and will discuss the individuals physical and emotional condition, current exercise level, accomplishment of previously set goals and action plans, and perceived barriers to participation in exercise. The assessor will use facilitation strategies to aid participants in devising strategies to overcome barriers and set realistic goals and action plans.
  Arms: Institution-Based Exercise and Self-Management (EXSM); Institution-Based Self-management only (SM)

SUMMARY:
BACKGROUND:

One in eight women will develop breast cancer in their lifetime. With improved screening and treatment techniques, more women are surviving breast cancer. However, women live with physical and emotional side effects secondary to treatment for years after cancer treatments have ended. Exercise can help to manage these side effects, however, less than 30% of this population takes part in regular exercise. The objective of this trial is to determine the feasibility and effectiveness of a novel exercise and education program for women with breast cancer during chemotherapy.

METHODS:

Participants in this study include women with a diagnosis of stage 1 - 3 breast cancer undergoing chemotherapy. Women will be divided into three groups. The first group will include 8 sessions of exercise and self-management education during their chemotherapy treatment. The second group will receive self-management education only, and the third group will receive usual care. Outcomes will be compared between groups at baseline, post-intervention, and at 6- and 12- month follow up. Outcomes to be assessed include exercise level, functional mobility, muscle strength, quality of life, health status, and use of health care services.

EXPECTED OUTCOMES:

Women with breast cancer are among the least active segment of the Canadian population. It is well known that inactivity can lead to physical and psychological side effects, cancer recurrence, and an increase in comorbid conditions. This proposed project addresses a long-standing need to help women with breast cancer become and stay more active by implementing a novel exercise and education program.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling
* English-speaking women
* over 18 years of age
* currently undergoing adjuvant or neoadjuvant chemotherapy for Stage 1-3 breast cancer
* cleared by their oncologist to participate in moderate intensity aerobic exercise

Exclusion Criteria:

* self-report any chronic condition, cognitive impairment, or injury that would prevent them from participating independently in moderate intensity exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change in baseline physical activity level | 16-weeks, 6-months, 12-months
  To be assessed using the Godin Leisure Time Exercise Questionnaire (total score 0-no maximum; higher scores indicating higher levels of physical activity) and activity tracker (Fitbit) data (demonstrating steps/day and total time of moderate levels of physical activity; higher scores indicate higher levels of activity).

SECONDARY OUTCOMES:
Change in baseline quality of life | 16-weeks, 6-months, 12-months
  Measured using the Functional Assessment of Cancer Therapy-Breast (measure of quality of life in breast cancer survivors; scale range 0-144; higher scores indicate higher levels of quality of life).
Change in level of exercise knowledge | 16-weeks, 6-months, 12-months
  Measured using the Theory of Planned Behaviour (TPB) based questionnaire (scale range 7-56; higher scores indicate higher levels of exercise knowledge).
Change in baseline perception of health status | 16-weeks, 6-months, 12-months
  Measured using the EQ-5D-3L a measure of health status (has two systems; a 3 level scale assessing five dimensions of health and a visual analogue scale from 0-10; higher scores indicate higher perceptions of health status)
Change in baseline aerobic capacity | 16-weeks, 6-months, 12-months
  Measured using the Six-minute walk test (6MWT) (a performance based measure that assesses total distance walked in six minutes, higher scores indicate higher levels of aerobic capacity)
Change in baseline levels of lower extremity strength | 16-weeks, 6-months, 12-months
  Measured using a manual muscle dynamometer (Movements assessed will be isometric hip and knee flexion/extension and ankle plantar flexion/dorsiflexion; higher scores indicate higher levels of lower extremity strength).
Change in patient engagement in health services | 16-weeks, 6-months, 12-months
  Measured using the Patient Health Engagement Scale (assesses five domains related to the experiences and preferences of patients for their engagement with their health care treatment; score range from 5-35; higher scores indicate higher levels of patient engagement in health services).
Change in baseline levels of resting BP | 16-weeks, 6-months, 12-months
  To measure change in cardiovascular outcomes; Measured with sphygmamometer
Change in baseline resting heart rate | 16-weeks, 6-months, 12-months
  To measure change in cardiovascular outcomes; Measured with pulsed oximeter

OTHER OUTCOMES:
Recruitment rate | At recruitment completion (approximately 1 year).
  Percentage of eligible patients actually enrolled in the study.
Retention rate | At intervention completion (Approximately 1.3 years).
  Percentage of enrolled patients who complete the intervention.
Drop out rate throughout study | At study completion (2 years)
  Percentage of participants who drop out from study at any time.
Representativeness of study sample | At recruitment completion (approximately 1 year).
  Descriptive characteristics of study samples (in regard to characteristics such as age, stage of cancer, fitness level, socio-economic status, etc.)
Adherence rate to intervention | At intervention completion (Approximately 1.3 years)
  Percentage of total intervention sessions attended.

CONTACTS AND LOCATIONS:
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith-Turchyn J, Mukherjee S, Richardson J, Ball E, Bordeleau L, Neil-Sztramko S, Levine O, Thabane L, Sathiyapalan A, Sabiston C. Evaluation of a novel strategy to implement exercise evidence into clinical practice in breast cancer care: protocol for the NEXT-BRCA randomised controlled trial. BMJ Open Sport Exerc Med. 2020 Oct 7;6(1):e000922. doi: 10.1136/bmjsem-2020-000922. eCollection 2020. PMID 33178447